CLINICAL TRIAL: NCT03522363
Title: Study of Streptococcus Dentisani Capacity to Colonize Supragingival Plaque in a Split Mouth Model
Brief Title: Streptococcus Dentisani Colonization Capacity in a Split Mouth Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ABB-Sdentcolonization
Record Dates: First submitted 2018-02-09; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-02

CONDITIONS: Oral Health
Keywords: oral health; Streptococcus dentisani

STUDY DESIGN:
Intervention Model Description: Phase I, exploratory, prospective, mechanistic pilot clinical trial with two parallel follow-up groups that differ in the number of treament applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monodose group (Experimental): 1 vial with 4E10 CFU/g Total dose treatment: 4E10 CFU
  Interventions: Other: Streptococcus dentisani CECT7746
- Multidose group (Experimental): 7 vials with 5,5E09 CFU/g Total dose treatment: 4E10 CFU
  Interventions: Other: Streptococcus dentisani CECT7746

INTERVENTIONS:
Other: Streptococcus dentisani CECT7746 — Treatment will be applied topically as an adhesive gel with a dental splint

SUMMARY:
Pilot study with healthy subjects to test the in vivo potential colonization ability of S. dentisani. Phase I, exploratory, prospective, mechanistic pilot clinical trial with two parallel follow-up groups. Probiotic will be applied topically as an adhesive gel with a dental splint under different dosing regimes. Saliva and plaque samples will be obtained at day 0, 14 and 28.

DETAILED DESCRIPTION:
Phase I study, exploratory, prospective, mechanistic, to evaluate the capacity of

Streptococcus dentisani CECT 7746 of colonizing the tooth surface. The study will be carried out with 10 healthy subjects divided into two groups (n = 5 per group) that differ in the number of applications of probiotic:

Group A: participants who will receive a single application of the product during the initial visit Group B: participants who will receive 7 applications on consecutive days, with the first in the start visit. Probiotic will be applied topically as an adhesive gel with a dental splint under different dosing regimes.The total dose received will be the same for both groups, and the total duration of the follow-up will be of 4 weeks from the first application also for both groups.

On day 0: Participants who meet the inclusion and exclusion criteria will be randomized in one of the two groups. Saliva and plaque samples will be obtained by the dentist, and all the participants will receive an professional teeth cleaning in one half of the mouth (quadrants 1-4). Afterwads, treatment will be applied by the dentist according to assigned group, and the randomized participants in the multiple-dose group will be explained how to perform the six successive applications at home every 24 hours.

On day 14: follow-up visit, saliva and plaque samples will be obtained from all participants. Patient assigned to the multi-dose group will return the used material On day 28th: final visit, saliva and plaque samples will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Absence of serious periodontal diseases (eg gingivitis, periodontitis)
* Ability to understand the requirements and implications of the study

Exclusion Criteria:

* Antibiotic consumption during the 30 days prior to the initiation of the study.
* Oral probiotics consumption during the 30 days before the start of the study
* Pregnant or lactating women
* Chronic diseases (eg, diabetes, kidney problems, cancer) or diseases that could affect salivary flow.
* Chronic treatment or medication that could reduce salivary flow, such as antidepressants or psychotropic drugs.
* Allergy to any of the product composition ingredients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
Streptococcus dentisani CECT 7746 colonization capacity | A measure to see the change in the Baseline Streptococcus dentisani adherence will be made in V1 and V2 (14 days and 28 days after the treatment beginning, respectivetly)
  Demonstrate the ability of Streptococcus dentisani CECT 7746 to adhere, colonize and remain in the dental surface after its application, with or without previous professional oral cleaning

SECONDARY OUTCOMES:
Streptococcus mutans concentration | 0 - 14- 28 days
  To evaluate if the administration of the probiotic S. dentisani CECT 7746 reduces the amount of oral Streptococcus mutans.
Oral acid production | 0 - 14- 28 days
  To evaluate if the administration of the S. dentisani CECT 7746 reduces the amount of acid produced after an oral sugar solution administration

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mira, Dr., Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Lluis Alcanyis Foundation dental clinic, University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided